CLINICAL TRIAL: NCT04289259
Title: National Real-life Study of Tumor Mutational Burden Assessment in First-line Lung Cancer
Brief Title: Tumor Mutational Burden in Lung Cancer Patients
Acronym: MUBULUC
Status: Terminated | Type: Observational
Why Stopped: The funder stopped to fund this study.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP180023; 2019-A00129-48 (Other: Agence nationale de sécurité du médicament et des produits de santé (French Competent Authority)); CA209-8RK (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Non Small Cell Lung Cancer; Non-Small Cell Carcinoma of Lung; Non Small Cell Lung Cancer Stage III; Non-small Cell Lung Cancer Stage IV
Keywords: Tumor mutational burden; Cancer gene panel; Whole-exome sequencing; FoundationOne CDx assay panel; RNA-sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 ml of blood samples will be collected to reach 10 ml of plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biopsy sample: Tumor mutational burden (TMB) will be assessed on a sample of the biopsy done during standard care of patients.
  Interventions: Other: TMB assessment
- Surgical sample: TMB will be assessed on a sample of the tumor surgical specimen resected during standard care of patients.
  Interventions: Other: TMB assessment
- Biopsy sample + surgical sample: TMB will be assessed both on a sample of the biopsy and a sample of the tumor surgical specimen resected during standard care of patients.
  Interventions: Other: TMB assessment

INTERVENTIONS:
Other: TMB assessment — Tumor mutational burden could be calculated by cancer gene panel (CGP), whole-exome sequencing (WES), RNA-sequencing (RNA-seq), FoundationOne CDx assay panel (FMI).

SUMMARY:
Tumor mutational burden (TMB) seems to be is an important marker for immune checkpoint inhibitors efficacy. This study aims to assess the feasibility of the TMB assessment in first-line lung cancer in routine practice both on biopsy and surgical tumor samples. Results will be an element of discussion for the generalization of the TMB implementation in cancer centers.

DETAILED DESCRIPTION:
1. Current knowledge about the field under investigation

   Clinical evidence demonstrates that treatment with immune checkpoint blocker (ICB) agents benefit to patients across multiple tumor type. However, development of predictive biomarkers is needed to identify patients who are most likely to respond to immunotherapy.

   An emerging biomarker for response to immunotherapy is the total number of mutations present in a tumor specimen. This biomarker is named mutation load or tumor mutational burden (TMB). It is hypothesized that highly mutated tumors are more likely to harbor neoantigens targeted by activated immune cells. This metric, allowed by recent advances in next-generation sequencing (NGS) technologies, notably whole-exome sequencing (WES) and RNA-sequencing (RNA-seq), has been shown, in several tumor types, to correlate with patient response to ICB. Indeed, the TMB has been correlated with clinical benefits of anti-PD-1 and anti-CTLA-4 therapy in various tumor types, including malignant melanoma (Snyder et al., 2014; Van Allen et al., 2015) with a threshold of more than 100 nonsynonymous single-nucleotide variants (nsSNV) per exome, non-small cell lung cancers (NSCLC) (Rizvi et al., 2015) with a threshold defined as superior to 178 nsSNVs per exome, and several DNA repair-deficient tumors (Howitt et al., 2015; Le et al., 2015, 2017). A recent study prospectively confirmed that the PFS among patients with a high tumor mutational burden was significantly longer with nivolumab plus ipilimumab than with chemotherapy in NSCLC (Hellmann et al., 2018). Overall, a direct link between DNA repair deficiency, mutational landscape, predicted neoantigen load, and clinical activity of ICB is suggested.

   TMB was defined as the number of somatic, coding, base substitution, and indel mutations per megabase of genome examined. All base substitutions and indels in the coding region of targeted genes. It has been shown that TMB calculated using cancer gene panel (CGP) assay agrees well with whole exome measures of mutation burden (Chalmers et al., 2017). This indicates that CGP, targeting the entire coding region of several hundred genes, covers sufficient genomic size to accurately assess WES mutational burden. It was found that filtering out germline alterations and rare variants was important to obtaining accurate measurements of TMB, and this will especially be important in patients from ethnic backgrounds not well represented in sequencing datasets. These findings indicate that CGP is an accurate, cost-effective, and clinically available tool for measuring TMB. The results of down sampling analysis show that the variation in measurement due to sampling when sequencing 1.1 Mb is acceptably low, resulting in highly accurate calling of TMB at a range of TMB levels. This sampling variation increases as the number of megabases sequenced decreases, especially at lower levels of TMB. While targeted CGP can be used to accurately assess TMB, it is not currently suited for identification of neoantigens, which might occur in any gene. Nevertheless, the theragnostic impact of TMB has been also determined with a targeted CGP by the FoundationOne CDx assay (Hellmann et al., 2018).

   The failure to assess the TMB may occur at different steps in the analytical process. It can be at the sample acquisition with a low level of DNA (5-10%). The NGS processing depending on the method can lead to a process failure around 2-3%. And finally, the bioinformatic curation will lead to a 3-5% of failure. At the end, the TMB will be undetermined with an attrition rate at 15% of the samples (Fondation Medicine Personal communication).

   The implementation of tumor mutational burden assessment in a nation-wide perspective is challenging and large efforts should be done. Whatever the method, WES or large CGP, the measurements of TMB will change the scale of gene sequencing in the molecular platforms.

   It is important that the platforms, where the tumor mutational burden measurement will be implemented can be able to calibrate their CGP and compared it to a standard reference for the measurement of TMB. Moreover, with the limited quantity of DNA, the implemented method needs to produce reliable result for most of the samples. The platforms need also to deploy their wet benches processes and their bioinformatics pipeline to be able to produce the TMB in a turnaround time compatible with clinical patients management.
2. Description of the population of study participants and justification for the choice of participants

   As mentioned above the TMB seems to be is an important marker for ICB efficacy. It is therefore important to implement the TMB measurement at a nationwide level to assure the equal access to the ICB.

   The French National Cancer Institute (INCa) has labelled molecular platforms which are in charge of the different molecular tests should establish their processes to be able to face to this new test. This study is designated to test different CGP methods to assess tumor mutational burden in lung cancers in order to compare the different methods and to identify the drawbacks and failures of the different methods. Results of this study should allow to estimate the needs for the implementation of TMB at the nationwide level, recommend cancer gene panels, propose validated bioinformatics pipelines and finally recommend preanalytical processes for reducing the failure rate of the tests.

   For this purpose this study will determine the TMB on patients with a lung cancer. 200 patients with a non-small cell lung cancer (NSCLC) and naive of treatment will be recruited.

   Three cohorts will be recruited:
   * 100 patients will be included without resection and we will determine the TMB on the biopsy specimen
   * 100 patients will be included after surgical resection of their tumor and we will determine the TMB on the resected specimen

     * Within this cohort, TMB will be assessed both on the biopsy specimen and on the resected specimen for 20 patients 200 patients will be enrolled in order to perform 220 TMB analysis.

   Participating sites are large platforms which were selected on the basis of their capacity to implement new tests and which have all facilities for conducting the described research. The patients included in this study will correspond to those that will receive immune checkpoint inhibitors during the course of their disease. This study in a non-interventional study, as it will not modify the clinical care of the patients. The tissue sampling will be taken during clinical procedure needed for patient care. The study will be proposed to patients after the verification that tissues have been collected in a way that is compatible with the present study. Only tumor material and no germline DNA will be collected.

   Selected patients will be close to those that receive ICB and the target population will be enriched with patients who had been surgically resected, in order to be able to have enough tissues to compare in these samples different methods to assess TMB and also to compare pre surgical biopsies and surgical specimen.
3. Description of the element or elements under investigation

Elements under investigation are the TMB of NSCLC patients. The attrition rate (number of cases without result) in the TMB estimation will be assessed. The gold standard for the determination of TMB is the WES as it covers all coding regions. Several others Cancer Gene Panel methods (CGP) have been described based on cancer gene panels sequencing. The CGP included in this study will be the panel from Illumina (TS500), Thermofisher (Oncomine Tumor Mutation Load Assay), home-made panel with Agilent technology (Dedicated XT HS) and Foundation medicine F1 CDx. It is recognized that size of the cancer gene panels should be close to 1Mb to be able to measure reliably the TMB in different type of cancer.

Different methods of measurement of TMB will be compared in this series on NSCLC in order to validate different CGP available on the market or in the different INCa platforms. Bioinformatics modelling will try to correlate the TMB results from WES and CGP. For this purpose, based on results of mutational load calculated from results of WES, results of mutation load will be extrapolated based on a random selection of 1000 genes repeated 1000 times. The mean of the correlation coefficient (R2) between the tumor mutational burden calculated by the whole exome sequencing and by the different random gene panels is 0.88 IQR [0.84-0.91] showing that the selection of genes to estimate the TMB should be evaluated carefully before to be used in clinical practice (unpublished results). The material that will be collected during the study will allow to determine the performance of the CGP implemented in the molecular biology platforms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with any NSCLC, stage III and IV with a molecular analysis on the French platform. There will be no exclusion criteria on the presence of an oncogenic mutation as EGFR, KRAS, ALK.
* Patient age will be ≥ 18 years old and < 85 years old
* The pre-analytical features of the patient's sample are compatible with the CGP / WES analysis.
* Patient has signed the ICF.
* The FFPE material from the patient's sample needs to be available to be analyzed on site and sent for central analyses. If FFPE sample is not available within 1 month, on-site analysis can begin on extracted DNA previously screened in small panel NGS.
* The neoplastic cells in the patient's sample should be superior to 30%.

Exclusion Criteria:

* The TMB in patient's NSCLC is already known or estimated in the case of a clinical trial.
* Patient with relapsing NSCLC if the initial cancer has received a neoadjuvant / adjuvant treatment.
* Patient under legal protection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a non-small cell lung cancer (NSCLC) and naive of treatment
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Global attrition rate | Time of sample analysis
  Number of cases without result

SECONDARY OUTCOMES:
Turnaround time to determine tumor mutational burden (TMB) | 3 weeks
  Time between the reception of the tissues samples on platforms and TMB results availability
Attrition rate for RNA-sequencing (RNAseq) | Time of sample analysis
  Number of cases analyzed by RNAseq approach without result
Rate of misclassification for TMB determined by RNA-seq | Time of sample analysis
  Compared to the TMB determined by whole exome sequencing (WES) as a gold standard
Rate of misclassification for TMB determined by Cancer Genome Panel (CGP) | Time of sample analysis
  Compared to the TMB determined by whole exome sequencing (WES) as a gold standard
Rate of misclassification for TMB determined by FoundationOne CDx assay panel | Time of sample analysis
  Compared to the TMB determined by whole exome sequencing (WES) as a gold standard
Molecular druggable alterations detected by CPG or WES and RNAseq | Time of sample analysis
Concordance of the TMB value in pre-surgical biopsies to surgical specimen for the same patients | Time of sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Cadranel, MD, Principal Investigator — AP-HP - Hôpital Tenon; Benjamin Besse, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Pierre Laurent-Puig, MD, Study Director — AP-HP - Hôpital Européen Georges-Pompidou; Etienne Rouleau, PharmD, PhD, Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (8):
- France (8):
  - Centre Jean Perrin, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Institut Bergonié, Bordeaux, Nouvelle-Aquitaine
  - Institut Curie, Paris, Île-de-France Region
  - AP-HP - Hôpital Cochin, Paris, Île-de-France Region
  - AP-HP - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region
  - AP-HP - Hôpital Tenon, Paris, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared.
  IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.